CLINICAL TRIAL: NCT00634088
Title: Parallel Phase I Study of Ixabepilone Plus Lapatinib and Ixabepilone Plus Lapatinib Plus Capecitabine in Subjects With HER2 Positive Locally Advanced or Metastatic Breast Cancer
Brief Title: Phase I Study of Ixabepilone Plus Lapatinib With or Without Capecitabine in the Treatment of Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual
Sponsor: R-Pharm (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA163-144; EURDRACT: 2007-004123-38
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Results first posted 2011-05-03 (Estimated); Last update posted 2016-03-10 (Estimated); Status verified 2016-02

CONDITIONS: Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Lapatinib; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg (Experimental): Dose Level 1
  Interventions: Drug: Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg (Experimental): Dose Level 2
  Interventions: Drug: Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg
- Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg (Experimental): Dose Level 3
  Interventions: Drug: Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg
- Ixabepilone + Lapatinib + Capecitabine (Experimental): Triplet Combination
  Interventions: Drug: Ixabepilone + Lapatinib + Capecitabine

INTERVENTIONS:
Drug: Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg — Lapatinib, 1000 mg, administered orally, once a day, every day, for 7 to 14 consecutive days as a lead-in period prior to the first administration of ixabepilone (Day 1). Following the lapatinib lead-in phase of Cycle 1, and on Day 1 of subsequent cycles, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1000 mg, administered orally, once a day, every day, for a 21-day cycle.
  Arms: Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg
Drug: Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg — Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1000 mg). Lapatinib, 1250 mg, administered orally once a day, every day, for 7 to 14 consecutive days as a lead-in period prior to the first administration of ixabepilone. Following the lapatinib lead-in phase of Cycle 1, and on Day 1 of subsequent cycles, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib administered, 1250 mg, orally, once a day, every day, for a 21-day cycle.
  Arms: Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg
Drug: Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg — Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1250 mg). Lapatinib, 1250 mg, administered orally once a day, every day, for 7 to 14 consecutive days as a lead-in period prior to the first administration of ixabepilone. Following the lapatinib lead-in phase of Cycle 1, and on Day 1 of subsequent cycles, ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1250 mg, administered orally, once a day, every day, for a 21-day cycle.
  Arms: Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg
Drug: Ixabepilone + Lapatinib + Capecitabine — Planned escalating doses of the triplet combination of ixabepilone, lapatinib, and capecitabine. No participants were enrolled in this arm due to premature termination of the study.
  Arms: Ixabepilone + Lapatinib + Capecitabine

SUMMARY:
The purpose of this study is to determine the safety and preliminary effectiveness of ixabepilone plus lapatinib with and without capecitabine in the treatment of human epidermal growth factor receptor 2 (HER2)-positive or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older with histologic or cytologic diagnosis of adenocarcinoma originating in the breast
* Radiologic or pathologic evidence that the cancer is metastatic or locally advanced (a T4 tumor and stage IIIB/IIIC disease) and not curable by local measures, such as radiation or surgery
* Positive status for human epidermal growth factor receptor 2
* Measurable disease as per Response Evaluation Criteria In Solid Tumors guidelines
* Karnofsky performance status of 70 to 100
* Life expectancy of at least 3 months

Exclusion Criteria:

* Prior radiation must not have included 30% or more of major bone-marrow containing areas, such as the pelvis and lumbar spine
* Common Terminology Criteria Grade 2 or greater neuropathy
* Inadequate hematologic, hepatic, or renal function
* Known prior severe hypersensitivity reactions to agents containing Cremophor® EL or known hypersensitivity or prior intolerance to fluoropyrimidine
* Known or suspected dihydropyrimidine dehydrogenase deficiency
* More than 3 prior chemotherapy regimens in the metastatic setting
* Prior treatment with an epothilone or lapatinib; prior treatment with capecitabine within the past 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (3):
- The Cancer Institute Of New Jersey, New Brunswick, New Jersey, United States
- Local Institution, Brisbane, Queensland, Australia
- Local Institution, Modena, Italy

REFERENCES:
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 13 participants enrolled, 10 received treatment with ixabepilone + lapatinib in escalating-dose cohorts. No participants were enrolled in the ixabepilone + lapatinib + capecitabine cohort due to premature termination of the study.
Groups:
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg: Lapatinib, 1000 mg, administered daily in a lead-in period, orally once a day, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib administered daily, orally once a day, for 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg: Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1000 mg). Lapatinib, 1250 mg, administered daily, orally once a day, for 7 to 14 consecutive days prior to the first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib administered daily, orally once a day, for 21-day cycle.
- Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg: Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1250 mg). Lapatinib, 1250 mg, administered daily, orally once a day, for 7 to 14 consecutive days prior to the first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion. Lapatinib administered daily, orally once a day, for 21-day cycle.
- Ixabepilone+ Lapatinib + Capecitabine: A triplet combination of ixabepilone, lapatinib, and capecitabine was planned for analysis in escalating doses but was not initiated due to premature termination of the study.
Period: Time Period 1: Dose Level 1
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone+ Lapatinib + Capecitabine
Started | 6 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 6 | 0 | 0 | 0
Not completed — Disease progression | 2 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0
Not completed — Adverse Event | 3 | 0 | 0 | 0
Period: Time Period 2: Dose Level 2
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone+ Lapatinib + Capecitabine
Started | 0 | 3 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 2 | 0 | 0
Not completed — Progressive disease | 0 | 1 | 0 | 0
Period: Time Period 3: Dose Level 3
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone+ Lapatinib + Capecitabine
Started | 0 | 0 | 1 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 1 | 0
Not completed — Progressive disease | 0 | 0 | 1 | 0
Period: Time Period 4: Triplet Combination
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone+ Lapatinib + Capecitabine
Started | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg: Lapatinib administered daily in escalating cohorts, beginning with 1000 mg, orally once a day, for 7 to 14 consecutive days in Cycle 1 prior to the first administration of ixabepilone. Then lapatinib administered daily, orally once a day, for a 21-day cycle. After the lapatinib lead-in phase, ixabepilone administered as a 3-hour IV infusion in escalating doses, beginning with 32 mg/m^2.
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg: Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1000 mg), lapatinib 1250 mg administered orally once a day, every day, for 7 to 14 consecutive days prior to the first administration of ixabepilone. Then lapatinib administered orally once a day, every day, for a 21-day cycle. After lapatinib lead-in period, ixabepilone administered as a 3-hour IV infusion of 32 mg/m^2.
- Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg: Initiated a minimum of 14 days following Day 1 of previous cohort (ixabepilone, 32 mg/m^2 + lapatinib, 1250 mg), lapatinib 1250 mg administered orally once a day, every day for 7 to 14 consecutive days prior to the first administration of ixabepilone in Cycle 1. Then lapatinib administered daily, orally once a day, for a 21-day cycle. Ixabepilone administered as a 3-hour IV infusion of 40 mg/m^2 following lapatinib lead-in period.
- Ixabepilone + Lapatinib + Capecitabine: A triplet combination of ixabepilone, lapatinib, and capecitabine was planned for analysis in escalating doses but was not initiated due to premature termination of the study.
- Total: Total of all reporting groups
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg | Ixabepilone + Lapatinib + Capecitabine | Total
Number analyzed (Participants) | 6 | 3 | 1 | 0 | 10
Age, Customized [Number; unit: participants]
  Younger than 50 years | 1 | 1 | 0 |  | 2
  50 years and older to younger than 65 years | 4 | 2 | 1 |  | 7
  65 years and older | 1 | 0 | 0 |  | 1
Gender [Number; unit: participants]
  Female | 6 | 3 | 1 |  | 10
  Male | 0 | 0 | 0 |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0 |  | 0
  Asian | 1 | 0 | 0 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 |  | 0
  Black or African American | 0 | 0 | 0 |  | 0
  White | 5 | 3 | 1 |  | 9
  More than one race | 0 | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) and Recommended Phase II Dose (RP2D) of Ixabepilone When Administered With Lapatinib
Description: The MTD is defined as the maximum dose that can be administered to 6 participants such that no more than 1 (or fewer than one third if more than 6 participants receive treatment) experiences a dose-limiting toxicity (DLT), with at least 2 experiencing a DLT at the next higher dose level. The RP2D is based on the MTD and the assessment of any relevant chronic toxicities.
Time Frame: Days 1 through 21
Population: Because the study was terminated due to insufficient enrollment, MTD was not achieved.
Groups:
- All Treated: All participants who received at least 1 dose of ixabepilone or lapatinib.
Arm/Group | All Treated
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) Leading to Discontinuation, Treatment-related AEs, Treatment-related AEs (Grade 3 or 4), Peripheral Neuropathy (PN), PN (Grade 3 or 4)
Description: AE=Any new untoward medical event or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. SAE=any untoward medical event that results in death, persistent or significant disability/incapacity, drug dependency or abuse; is life-threatening, important, a congenital anomaly/birth defect; or requires or prolongs existing hospitalization. Treatment related=possibly, probably, or certainly related to and of unknown relationship to study treatment. Common Terminology Criteria (CTC) Grade 3=severe; Grade 4=life-threatening or disabling.
Time Frame: Baseline to Day 21, continuously
Population: All participants who received at least 1 dose of ixabepilone and either lapatinib or capecitabine.
Measure: Number; unit: Participants
Groups:
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d: Lapatinib, 1000 mg, administered daily, orally once a day, at least 1 hour before or after a meal, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase of Cycle 1, and on Day 1 of subsequent cycles, ixabepilone, 32 mg/m^2, administered as a 3-hour intravenous (IV) infusion. Lapatinib, 1000 mg, administered daily, orally once a day, for a 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d: Lapatinib, 1250 mg, administered daily, orally once a day, at least 1 hour before or after a meal, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase of Cycle 1 and on Day 1 of subsequent cycles, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1250 mg, administered daily, orally once a day, for a 21-day cycle.
- Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d: Lapatinib, 1250 mg, administered daily, orally once a day, at least 1 hour before or after a meal, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase of Cycle 1, and on Day 1 of subsequent cycles, ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1250 mg, administered daily, orally once a day, for a 21-day cycle.
- Ixabepilone + Lapatinib + Capecitabine: Planned escalating doses of ixabepilone, 32 to 40 mg/m^2 + lapatinib, 1000 to 1250 mg + capecitabine, 1650 to 2000 mg/m^2. No participants were enrolled in this arm due to premature termination of the study.
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 6 | 3 | 1 | 0
Participants
  Death | 3 | 0 | 0 |
  SAEs | 2 | 0 | 1 |
  AEs leading to discontinuation | 3 | 2 | 0 |
  Treatment-related AEs | 6 | 3 | 1 |
  Treatment-related AEs (Grade 3 or 4) | 3 | 3 | 1 |
  PN | 4 | 2 | 0 |
  PN (Grade 3 or 4) | 1 | 1 | 0 |

3. Secondary Outcome: Number of Participants With DLT
Description: DLT=Any of the following events, attributable to study drug and occurring within 21 days after ixabepilone administration: Grade 3 or 4 nausea, vomiting, or diarrhea despite the use of adequate medical intervention; other Grade 3 or greater nonhematologic toxicity requiring removal from study drug; recovery from study drug-related toxicity that delayed scheduled retreatment for longer than 3 weeks; Grade 4 neutropenia for 5 or more consecutive days or Grade 3 or 4 neutropenia of any duration with sepsis or fever; thrombocytopenia or bleeding requiring platelet transfusion.
Time Frame: Baseline to Day 21, continuously
Population: All participants who received at least 1 dose of ixabepilone and either lapatinib or capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 6 | 3 | 1 | 0
Participants | 1 | 0 | 0 |

4. Secondary Outcome: Number of Participants With Abnormalities in Hematology Laboratory Results by Worst CTC Grade
Description: CTC, Version 3.0 used to assess parameters. ULN=upper level of normal among all laboratory ranges. WBC (c/L): Grade (Gr)1:<LLN to 3.0*10^9/L, Gr 2:<3.0 to 2.0*10^9/L, Gr 3:<2.0 to 1.0*10^9/L, Gr 4:<1.0*10^9/L; ANC (c/uL): Gr 1:<LLN to 1.5*10^9/L, Gr 2:<1.5 to 1.0*10^9/L, Gr 3:<1.0 to 0.5*10^9/L, Gr 4:<0.5*10^9/L; Platelet count (c/uL): Gr 1:LLN to 75.0*10^9/L, Gr 2:<75.0 to 50.0*10^9/L, Gr 3:<50.0 to 25.0*10^9/L, Gr 4:<25.0*10^9/L; Hemoglobin (g/dL): Gr 1:<LLN to 10.0 g/dL, Gr 2:<10.0 to 8.0 g/dL, Gr 3:<8.0 to 6.5 g/dL, Gr 4:<6.5 g/dL.
Time Frame: Baseline and weekly from Days 1 to 21 (Cycle 1)
Population: All participants who received at least 1 dose of ixabepilone and either lapatinib or capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 6 | 3 | 1 | 0
Participants
  White blood cell count (WBC) (Grade 1) | 1 | 0 | 1 |
  WBC (Grade 2) | 1 | 0 | 0 |
  WBC (Grade 3) | 2 | 3 | 0 |
  WBC (Grade 4) | 1 | 0 | 0 |
  Absolute neutrophil count (ANC) (Grade 1) | 0 | 0 | 0 |
  ANC (Grade 2) | 1 | 0 | 0 |
  ANC (Grade 3) | 2 | 1 | 0 |
  ANC (Grade 4) | 2 | 2 | 0 |
  Platelet count (Grade 1) | 1 | 1 | 2 |
  Platelet count (Grade 2) | 0 | 0 | 0 |
  Platelet count (Grade 3) | 0 | 0 | 0 |
  Platelet count (Grade 4) | 0 | 0 | 0 |
  Hemoglobin (Grade 1) | 3 | 3 | 6 |
  Hemoglobin (Grade 2) | 3 | 0 | 4 |
  Hemoglobin (Grade 3) | 0 | 0 | 0 |
  Hemoglobin (Grade 4) | 0 | 0 | 0 |

5. Secondary Outcome: Number of Participants With Abnormalities in Serum Chemistry Laboratory Results by Worst CTC Grade
Description: CTC, Version 3.0 used to assess parameters. ULN=upper level of normal among all laboratory ranges. ALT(U/L) Gr 1:>ULN-2.5*ULN,Gr 2:>2.5-5.0*ULN,Gr 3:>5.0-20.0*ULN,Gr 4:>20.0* ULN; AST(U/L) Gr 1:>ULN-2.5* ULN,Gr 2:>2.5-5.0*ULN,Gr 3:>5.0-20.0*ULN,Gr 4:>20.0* ULN; ALP(U/L)Gr 1:>ULN-2.5*ULN, Gr 2:>2.5-5.0*ULN, Gr 3:>5.0-20.0*ULN, Gr 4:>20.0*ULN; Creatinine (mg/dL): Gr 1:>ULN-1.5*ULN, Gr 2:>1.5-3.0*ULN, Gr 3:>3.0-6.0*ULN, Gr 4:>6.0*ULN; Total bilirubin (mg/dL): Gr 1:>ULN-1.5*ULN, Gr 2:>1.5-3.0*ULN, Gr 3:>3.0-10.0*ULN, Gr 4:>10.0*ULN
Time Frame: At baseline and within 72 hours of Day 1 of 21-day cycle
Population: All participants who received at least 1 dose of ixabepilone and either lapatinib or capecitabine.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 6 | 3 | 1 | 0
Participants
  Alanine aminotransferase (ALT) (Grade 1) | 1 | 0 | 0 |
  ALT (Grade 2) | 0 | 0 | 0 |
  ALT (Grade 3) | 0 | 0 | 0 |
  ALT (Grade 4) | 0 | 0 | 0 |
  Aspartate aminotransferase (AST) (Grade 1) | 1 | 0 | 0 |
  AST (Grade 2) | 0 | 0 | 0 |
  AST (Grade 3) | 0 | 0 | 0 |
  AST (Grade 4) | 0 | 0 | 0 |
  Alkaline phosphatase (ALP) (Grade 1) | 3 | 0 | 0 |
  ALP (Grade 2) | 0 | 0 | 0 |
  ALP (Grade 3) | 0 | 0 | 0 |
  ALP (Grade 4) | 0 | 0 | 0 |
  Creatinine (Grade 1) | 0 | 0 | 0 |
  Creatinine (Grade 2) | 0 | 0 | 0 |
  Creatinine (Grade 3) | 0 | 0 | 0 |
  Creatinine (Grade 4) | 0 | 0 | 0 |
  Total bilirubin (Grade 1) | 0 | 0 | 0 |
  Total bilirubin (Grade 2) | 0 | 0 | 0 |
  Total bilirubin (Grade 3) | 0 | 0 | 0 |
  Total bilirubin (Grade 4) | 0 | 0 | 0 |

6. Secondary Outcome: Maximum Concentration of Ixabepilone
Time Frame: Day 1 of 21-day cycle
Population: Participants who received ixabepilone with lapatinib treatment and had pharmacokinetic parameters available.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 5 | 3 | 1 | 0
ng/mL | 200.6 (78.4) [105.5 to 311.1] | 109.2 (1.1) [107.9 to 110.1] | 133.4 [133.4 to 133.4] |

7. Secondary Outcome: Area Under the Concentration-time Curve From 0 to Infinity (AUC[INF]) and AUC From 0 to Last Quantifiable Concentration (AUC[O-T] of Ixabepilone
Time Frame: Day 1 of 21-day cycle
Population: Participants who received ixabepilone with lapatinib treatment and had pharmacokinetic parameters available.
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 5 | 3 | 1 | 0
ng*h/mL
  AUC(INF) | 2212.9 (1030.4) | 2427.0 (225.5) | 1610.7 |
  AUC(O-T) | 1851.8 (880.5) | 2082.0 (133.6) | 1284.2 |

8. Secondary Outcome: Terminal Half-life of Ixabepilone
Time Frame: Day 1 of 21-day cycle
Population: Participants who received ixabepilone with lapatinib treatment and had pharmacokinetic parameters available.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 5 | 3 | 1 | 0
Hours | 51.6 (13.2) | 63.1 (10.4) | 33.1 |

9. Secondary Outcome: Time to Peak Concentration of Ixabepilone
Time Frame: Day 1 of 21-day cycle
Population: Participants who received ixabepilone with lapatinib treatment and had pharmacokinetic parameters available.
Measure: Median (Full Range); unit: Hours
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 5 | 3 | 1 | 0
Hours | 3.0 [2.0 to 3.4] | 3.0 [3.0 to 3.0] | 2.9 [2.9 to 2.9] |

10. Secondary Outcome: Volume of Distribution at Steady State of Ixabepilone
Time Frame: Day 1 of 21-day cycle
Population: Participants who received ixabepilone with lapatinib treatment and had pharmacokinetic parameters available.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 5 | 3 | 1 | 0
Liters | 1484.3 (438.5) | 1780.8 (237.9) | 1915.8 |

11. Primary Outcome: MTD and RP2D of Ixabepilone When Administered With Lapatinib Plus Capecitabine
Description: MTD is defined as the maximum dose that can be administered to 6 participants such that no more than 1 (or fewer than one third if more than 6 participants receive treatment) experiences a DLT, with at least 2 experiencing a DLT at the next higher dose level. The RP2D is based on the MTD and the assessment of any relevant chronic toxicities.
Time Frame: Days 1 through 21
Population: Because the study was terminated due to insufficient enrollment, no participants received the triplet combination.
Arm/Group | All Treated
Number analyzed (Participants) | 0

12. Secondary Outcome: Overall Tumor Response By Number of Participants
Description: Target lesion criteria: Complete Response(CR)=Disappearance of all clinical and radiologic evidence of target lesions; Partial Response (PR)=A 30% or greater decrease in the sum of longest diameter(LD) of all lesions in reference to the baseline sum LD. Stable Disease (SD)=Insufficient increase to qualify for Progressive Disease (PD) and insufficient shrinkage to qualify for PR; PD=A 20% or greater increase in the sum of LD of all target lesions, taking as reference the smallest sum LD recorded at or following baseline.
Time Frame: Baseline and Day 21 (21-day cycle)
Population: All participants with measurable disease at baseline per RECIST guidelines, with the exception of those with an incorrect diagnosis.
Measure: Number; unit: Participants
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 6 | 3 | 1 | 0
Participants
  CR | 3 (12.2) | 2 (2.1) | 0 |
  PR | 0 | 0 | 0 |
  SD | 3 | 1 | 1 |
  PD | 0 | 0 | 0 |

13. Secondary Outcome: Duration of Response of Combination Treatment With Ixabepilone Plus Lapatinib
Description: Duration of response is measured from the time in months that measurement criteria are first met for PR or CR, whichever is recorded first, until the date of documented PD or death. Participants who neither relapse nor die will be censored on the date of their last tumor assessment.
Time Frame: First occurrence of PR or CR to PD or Death (no average, as no data available)
Population: Because the study was terminated due to insufficient enrollment, the duration of response could not be analyzed.
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone + Lapatinib + Capecitabine
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to Day 21, continuously
Groups:
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d: Lapatinib, 1000 mg, administered daily in a lead-in period, orally once a day, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1000 mg, administered daily, orally once a day, for 21-day cycle.
- Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d: Lapatinib, 1250 mg, administered daily in a lead-in period, orally once a day, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 32 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1250 mg, administered daily, orally once a day, for 21-day cycle.
- Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d: Lapatinib, 1250 mg, administered daily in a lead-in period, orally once a day, for 7 to 14 consecutive days prior to first administration of ixabepilone (Day 1). After the lapatinib lead-in phase, ixabepilone, 40 mg/m^2, administered as a 3-hour IV infusion. Lapatinib, 1250 mg, administered daily, orally once a day, for 21-day cycle.
Arm/Group | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d
Serious Adverse Events (participants affected / at risk) | 2/6 | 0/3 | 1/1
Other Adverse Events (participants affected / at risk) | 6/6 | 3/3 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d (N=6) | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d (N=3) | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d (N=1)
NAUSEA (Gastrointestinal disorders) | 0 | 0 | 1
VOMITING (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 | 0 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 | 0 | 0
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ixabepilone, 32 mg/m^2 + Lapatinib, 1000 mg/d (N=6) | Ixabepilone, 32 mg/m^2 + Lapatinib, 1250 mg/d (N=3) | Ixabepilone, 40 mg/m^2 + Lapatinib, 1250 mg/d (N=1)
CATARACT (Eye disorders) | 1 | 0 | 0
CYCLOPLEGIA (Eye disorders) | 1 | 0 | 0
VISION BLURRED (Eye disorders) | 1 | 0 | 0
VISUAL ACUITY REDUCED (Eye disorders) | 1 | 0 | 0
NEUROLOGICAL EYELID DISORDER (Eye disorders) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 1 | 0
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0 | 1
BLOOD MAGNESIUM DECREASED (Investigations) | 1 | 0 | 0
BLOOD POTASSIUM DECREASED (Investigations) | 2 | 0 | 0
EJECTION FRACTION DECREASED (Investigations) | 0 | 1 | 0
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 0 | 1 | 0
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 1 | 0 | 0
FLUSHING (Vascular disorders) | 1 | 0 | 0
LYMPHOEDEMA (Vascular disorders) | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 1 | 0 | 0
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 | 0 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 0 | 0
PORTAL VEIN THROMBOSIS (Hepatobiliary disorders) | 1 | 0 | 0
DRUG HYPERSENSITIVITY (Immune system disorders) | 2 | 0 | 0
AGEUSIA (Nervous system disorders) | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 2 | 0 | 0
LETHARGY (Nervous system disorders) | 1 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 1 | 1 | 0
NEURALGIA (Nervous system disorders) | 1 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 0 | 0
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 4 | 2 | 0
NAUSEA (Gastrointestinal disorders) | 5 | 1 | 1
VOMITING (Gastrointestinal disorders) | 3 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 5 | 3 | 1
GASTRITIS (Gastrointestinal disorders) | 0 | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 2 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 1 | 0 | 0
PARAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0
HYPOAESTHESIA ORAL (Gastrointestinal disorders) | 1 | 0 | 0
FAECAL INCONTINENCE (Gastrointestinal disorders) | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 1 | 0 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0
FOLLICULITIS (Infections and infestations) | 0 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 0
LOCALISED INFECTION (Infections and infestations) | 2 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 1
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 2 | 0 | 0
POLLAKIURIA (Renal and urinary disorders) | 1 | 0 | 0
MICTURITION URGENCY (Renal and urinary disorders) | 0 | 0 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 1
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 0 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2 | 0 | 1
ANAEMIA (Blood and lymphatic system disorders) | 2 | 0 | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 0 | 2 | 0
NEUTROPENIA (Blood and lymphatic system disorders) | 3 | 3 | 0
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 1 | 2 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
ONYCHOLYSIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PAIN OF SKIN (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
RASH MACULAR (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 2 | 1 | 0
HYPOAESTHESIA FACIAL (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 2 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 0 | 0
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PAIN (General disorders) | 1 | 0 | 0
FATIGUE (General disorders) | 4 | 1 | 0
PYREXIA (General disorders) | 1 | 0 | 0
EXTRAVASATION (General disorders) | 1 | 0 | 0
CHEST DISCOMFORT (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 3 | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period of 60 days or less from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.